CLINICAL TRIAL: NCT01659034
Title: Short and Optimal Duration of Dual Antiplatelet Therapy Study
Acronym: STOPDAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-645
Record Dates: First submitted 2012-07-30; First posted 2012-08-07 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: Anti-platelet therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — thienopyridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thienopyridine (Experimental): Thienopyridine treatment for 3 months after implantation of everolimus-eluting Stents
  Interventions: Drug: Thienopyridine for 3 months

INTERVENTIONS:
Drug: Thienopyridine for 3 months

SUMMARY:
The purpose of this study is to evaluate safety of reduction of thienopyridine treatment period to 3 months after implantation of Cobalt-Chromium everolimus-eluting Stents.

DETAILED DESCRIPTION:
"Thienopyridine antiplatelet agents have markedly inhibited incidence of stent thrombosis, when they were combined with aspirin for 1 month after implantation of bare-metal stent (BMS). On the other hand, combination of aspirin with thienopyridine (dual antiplatelet therapy: DAPT) for more than 1 year after drug-eluting stent (DES) implantation is frequently used to prevent very late stent thrombosis in the current clinical practice. In the RESET study, which was carried out in clinical practice in Japan, DAPT was performed for at least 1 year in 90% of the patients. However, there has been no report showing that long-term thienopyridine treatment for at least 1 year reduces incidence of serious cardiovascular events, and large-scale observational studies or small-scale randomized comparative studies have demonstrated that thienopyridine treatment for 6 months or for at least 12 months does not reduce incidence of serious cardiovascular events. These results suggest that the optimal duration of DAPT after DES implantation may be shorter than 6 months.

With respect to Everolimus-eluting stent (EES), which is the most widely used DES in Japan, it has been associated with significantly lower incidence of early or late stent thrombosis compared with the first-generation DES and with BMS in large-scale observational study and randomized comparative studies and their meta-analyses.

Considering that long-term DAPT obviously increases hemorrhagic complications compared to Aspirin monotherapy, it is desirable to reduce the duration of DAPT as far as possible, if long-term DAPT is not effective in inhibiting the incidence of serious cardiovascular events. Moreover, long-term DAPT enormously increases medical expenses. In this study, we planned an exploratory multicenter study to evaluate incidences of cardiovascular events and bleeding events at 12 months after stent implantation using an EES (XIENCE Prime™), which is associated with low risk of stent thrombosis, when thienopyridine therapy is discontinued at 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received PCI using everolimus-eluting cobalt-chromium stents

Exclusion Criteria:

* Patients who had been implanted drug-eluting stents other than everolimus-eluting cobalt-chromium stents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1525 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular and bleeding events | 1-year
  Composite of cardiovascular death, myocardial infarction, stroke (ischemic and hemorrhagic), stent thrombosis (definite stent thrombosis not resulting in myocardial infarction), and major bleeding (TIMI Major/Minor) Cardiovascular death, myocardial infarction and stent thrombosis are defined according to the definition in the Academic Research Consortium (ARC). Stroke is defined as ischemic or hemorrhagic stroke with symptoms lasting > 24 hour. Major bleeding is defined according to the definition in the Thrombosis in Myocardial Infarction (TIMI).

SECONDARY OUTCOMES:
Cardiovascular death/MI/stroke/definite ST | 1-year
  Composite of cardiovascular death, myocardial infarction, stroke, and definite stent thrombosis
Major bleeding (TIMI Major/Minor) | 1-year
  Major bleeding (TIMI Major/Minor)
Death/MI | 1-year
  Composite of all-cause death and myocardial infarction
All-cause death | 1-year
  All-cause death
Cardiovascular death/MI | 1-year
  Composite of cardiovascular death and myocardial infarction
Cardiovascular death | 1-year
  Cardiovascular death
MI | 1-year
  Myocardial infarction
Stroke | 1-year
  Both ischemic and hemorrhagic stroke excluding transient ischemic attack
Stent Thrombosis | 1-year
  Stent thrombosis according to Academic Research Consortium classification
Target Lesion Failure | 1-year
  Composite of cardiovascular death, myocardial infarction due to target vessel, and target lesion revascularization
Target Vessel Failure | 1-year
  Composite of cardiovascular death, myocardial infarction, and target vessel revascularization
Major Adverse Cardiac Events | 1-year
  Composite of cardiovascular death, myocardial infarction, and clinically-driven target lesion revascularization
Target Lesion Revascularization | 1-year
  Target lesion revascularization
Clinically-driven Target Lesion Revascularization | 1-year
  Clinically-driven Target Lesion Revascularization
Non Target Lesion Revascularization | 1-year
  Revascularization for non-target vessel or target vessel but target lesion
CABG | 1-year
  Coronary artery bypass graft
Target Vessel Revascularization | 1-year
  Target vessel revascularization
Any bleeding | 1-year
  Any bleeding complications

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Principal Investigator — Professor of Medicine, Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Department of Cardiovascular Medicine, Kyoto University Hospital, Kyoto, Kyoto, Japan